CLINICAL TRIAL: NCT00477672
Title: A Multi-Center, Placebo-Controlled, Double-Blind Trial to Examine the Safety and Efficacy of ACP-103 in the Treatment of Psychosis in Parkinson's Disease
Brief Title: A Study of the Safety and Efficacy of Pimavanserin (ACP-103) in Patients With Parkinson's Disease Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-012
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Parkinson's Disease Psychosis
Keywords: Parkinson's disease, psychotic disorders
MeSH Terms: conditions — Parkinson Disease; Psychotic Disorders | interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 (Experimental): Pimavanserin tartrate (ACP-103), 10 mg, tablet, once daily by mouth, 6 weeks
  Interventions: Drug: Pimavanserin tartrate (ACP-103)
- 3 (Experimental): Pimavanserin tartrate (ACP-103), 40 mg, tablet, once daily by mouth, 6 weeks
  Interventions: Drug: Pimavanserin tartrate (ACP-103)
- 1 (Placebo Comparator): Placebo tablet, once daily by mouth, 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimavanserin tartrate (ACP-103) — 10 mg, tablet, once daily by mouth, 6 weeks
  Arms: 2
Drug: Pimavanserin tartrate (ACP-103) — 40 mg, tablet, once daily by mouth, 6 weeks
  Arms: 3
Drug: Placebo — tablet, once daily by mouth, 6 weeks
  Arms: 1

SUMMARY:
This study will evaluate the safety and efficacy of two dose levels of pimavanserin (ACP-103) compared to placebo in patients with Parkinson's disease psychosis.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Parkinson's disease with a minimum duration of 1 year
* Presence of visual and/or auditory hallucinations, and/or delusions, occurring during the four weeks prior to study screening
* Psychotic symptoms must have developed after PD diagnosis was established
* Subject must be on stable dose of anti-Parkinson's medication for 1 month prior to Study Day 1 (Baseline) and during the trial
* Subject that has received stereotaxic surgery for subthalamic nucleus deep brain stimulation must be at least 6 months post surgery and the stimulator settings must have been stable for at least 1 month prior to Study Day 1 (Baseline) and must remain stable during the trial
* The subject is willing and able to provide consent
* Caregiver is willing and able to accompany the subject to all visits

Exclusion Criteria:

* Subject has a history of significant psychotic disorders prior to or concomitantly with the diagnosis of Parkinson's disease including, but not limited to, schizophrenia or bipolar disorder
* Subject has received previous ablative stereotaxic surgery (i.e., pallidotomy and thalamotomy) to treat Parkinson's disease
* Subject has current evidence of a serious and or unstable cardiovascular, respiratory, gastrointestinal, renal, hematologic or other medical disorder
* Subject has had a myocardial infarction in last six months
* Subject has any surgery planned during the screening, treatment or follow-up periods

Patients will be evaluated at screening to ensure that all criteria for study participation are met. These evaluations will include specific measures of psychosis severity, delirium, dementia, cardiovascular condition, and pregnancy status. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all protocol-specified entry criteria).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (36):
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Berkeley, California
  - Carson, California
  - Fountain Valley, California
  - Irvine, California
  - Sunnyvale, California
  - Danbury, Connecticut
  - Fairfield, Connecticut
  - Boca Raton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pompano Beach, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Springfield, Illinois
  - Scarborough, Maine
  - Worcester, Massachusetts
  - Southfield, Michigan
  - Traverse City, Michigan
  - Toms River, New Jersey
  - Kingston, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Salisbury, North Carolina
  - Columbus, Ohio
  - Warwick, Rhode Island
  - Brentwood, Tennessee
  - San Antonio, Texas
  - Richmond, Virginia
  - Kirkland, Washington
  - Spokane, Washington
- Bulgaria (4):
  - Pleven
  - Rousse
  - Sofia
  - Varna
- France (6):
  - Clermont-Ferrand
  - Marseille
  - Nantes
  - Pessac
  - Strasbourg
  - Toulouse
- India (9):
  - Bangalore
  - Hyderabad
  - Karnataka
  - Mangalore
  - Mumbai
  - New Dalhi
  - Pune
  - Tamil Nadu
  - Visakhapatnam
- Russia (6):
  - Kazan'
  - Kirov
  - Moscow
  - Saint Petersburg
  - Samara
  - Smolensk
- Ukraine (5):
  - Kharkiv
  - Kiev
  - Luhansk
  - Lviv
  - Vinnytsia
- United Kingdom (8):
  - Barnsley
  - Blackburn
  - Brighton
  - Dorset
  - London
  - Newcastle upon Tyne
  - North Shields
  - Salford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet, once daily by mouth, 6 weeks
- Pimavanserin 10 mg: Pimavanserin tartrate (ACP-103) 10 mg, tablet, once daily by mouth, 6 weeks
- Pimavanserin 40 mg: Pimavanserin tartrate (ACP-103) 40 mg, tablet, once daily by mouth, 6 weeks
Period: Overall Study
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 40 mg
Started | 98 | 101 | 99
Completed | 91 | 85 | 83
Not Completed | 7 | 16 | 16
Not completed — Adverse Event | 3 | 5 | 6
Not completed — Death | 0 | 1 | 0
Not completed — Disease progression | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol noncompliance | 0 | 2 | 0
Not completed — Consent withdrawn | 2 | 5 | 10
Not completed — Discretion of Sponsor | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 40 mg | Total
Number analyzed (Participants) | 98 | 99 | 98 | 295
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 30 | 23 | 80
  >=65 years | 71 | 69 | 75 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (9.67) | 69.0 (8.61) | 69.4 (7.84) | 69.3 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 36 | 24 | 107
  Male | 51 | 63 | 74 | 188
Region of Enrollment [Number; unit: participants]
  United States | 44 | 45 | 45 | 134
  India | 10 | 10 | 10 | 30
  Europe | 44 | 44 | 43 | 131

OUTCOME MEASURES:

1. Primary Outcome: Antipsychotic Efficacy
Description: Antipsychotic Efficacy was defined as a decrease in the severity and/or frequency of hallucinations and/or delusions. This is measured as the change from baseline (Day 1) to Day 42 in the Scale for the Assessment of Positive Symptoms - Hallucinations and Delusions scales (SAPS-H+D) score for the ITT Analysis Set. The possible total score is 0 to 100 and a negative change in score indicates improvement.
  Analysis Method: Analysis of Covariance (ANCOVA) and missing data was imputed using Last Observation Carried Forward (LOCF) method.
Time Frame: Each study visit (i.e. Days 1, 8, 15, 29 and 42)
Population: This is the "Intent to Treat" population, defined as patients who received at least one dose of study drug, and had both the baseline SAPS assessment and at least one post-baseline SAPS assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on the SAPS H+D scale
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 40 mg
Number analyzed (Participants) | 95 | 96 | 91
Score on the SAPS H+D scale
  Change from Baseline | -5.9 (7.90) [-7.3 to -4.5] | -5.8 (9.77) [-7.2 to -4.3] | -6.7 (7.87) [-8.1 to -5.2]
  Difference of Least Squares Mean versus Placebo | NA [NA to NA] — Calculation is a comparison of active arm versus placebo. | 0.1 [-1.7 to 2.0] | -0.8 [-2.7 to 1.1]

2. Secondary Outcome: Motor Symptoms Change From Baseline (Negative = Improvement)
Description: Motor symptoms were measured using the change from baseline (Day 1) to Day 42 in the combined score of the Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living) and Part III (Motor Examination) using the per-protocol (PP) analysis set. The possible total score is 0 to 160 and a negative change in score indicates improvement.
  Analysis Method: ANCOVA, and missing data was imputed using LOCF. The UPDRS Parts II+III score was analyzed by constructing 2-sided 95% confidence intervals (CIs) on the difference between each pimavanserin dose group and placebo mean change from baseline. Non-inferiority was concluded if the upper limit of the CI was less than or equal to 5.
Time Frame: Each study visit (i.e. Days 1, 8, 15, 29 and 42)
Population: This is the "Per Protocol" population, which includes subjects in the ITT analysis set, who were free of important protocol deviations, as defined before database lock and unblinding. Subjects were analyzed according to the treatment actually received.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on UPDRS-II+III
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 40 mg
Number analyzed (Participants) | 90 | 88 | 85
Score on UPDRS-II+III
  Change from Baseline | -2.94 [-5.08 to -0.80] | -1.41 [-3.58 to 0.76] | -3.13 [-5.34 to -0.91]
  Difference of Least Square Mean versus Placebo | NA [NA to NA] — Calculation is a comparison of active arm versus placebo. | 1.53 [-1.24 to 4.31] | -0.19 [-2.99 to 2.62]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: From the time the informed consent was signed, adverse events were recorded in the subject's source documents and entered into the appropriate eCRF pages at the Screening visit, at visits on Study Days 1, 8, 15, 29, 42 and Day 70 or 4 weeks after the last dose for subjects who do not continue into the open-label, extension protocol.
Arm/Group | Placebo | Pimavanserin 10 mg | Pimavanserin 40 mg
Serious Adverse Events (participants affected / at risk) | 2/98 | 5/99 | 5/98
Other Adverse Events (participants affected / at risk) | 34/98 | 29/99 | 27/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | Pimavanserin 10 mg (N=99) | Pimavanserin 40 mg (N=98)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dementia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=98) | Pimavanserin 10 mg (N=99) | Pimavanserin 40 mg (N=98)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (5) | 8 (10)
Constipation (Gastrointestinal disorders) | 3 (4) | 4 (5) | 5 (5)
Edema (General disorders) | 1 (1) | 2 (3) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 11 (12) | 5 (5) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4) | 7 (7) | 7 (7)
Headache (Nervous system disorders) | 6 (6) | 4 (4) | 4 (4)
Confusional state (Psychiatric disorders) | 3 (3) | 5 (5) | 5 (5)
Orthostatic hypotension (Vascular disorders) | 9 (10) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.